CLINICAL TRIAL: NCT06509503
Title: Impact of Combined Oral Contraceptive Pills on Migraine, a Randomized Controlled Trial
Brief Title: Impact of Combined Oral Contraceptive Pills on Migraine
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Sherihan Rezk Ahmed, principal investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 091287
Record Dates: First submitted 2024-07-13; First posted 2024-07-19 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Migraine
Keywords: migraine; combined oral contraception; Egypt
MeSH Terms: conditions — Migraine Disorders | interventions — Contraceptives, Oral, Combined; Contraceptive Devices, Female

STUDY DESIGN:
Intervention Model Description: We have two groups; the first group will include 200 patients who received COCs, while the second group will receive mechanical contraception We will assess the number of migraine days after three months of treatment and the percentage of patients who achieved ≥ 50% reduction in the monthly headache days frequency compared to the baseline frequency. HIT-6 score reduction in each group after three months of treatment. The safety of treatment was evaluated by monitoring and documenting treatment-emergent adverse events (TEAE) in patients through regular follow-up procedures for three months and the phenotypic features of migraine in each group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the COCs group (Active Comparator): The arm will include 200 migraine patients diagnosed according to ICHD3-beta criteria. The patients are regular users of COCs and will receive propranolol 80-160mg daily and ibuprofen 200-400 mg only in acute migraine attacks for 3 months. We will assess The change in migraine days per 28 days, the number of migraine days after three months of treatment, and the percentage of patients who achieved ≥ 50% reduction in the monthly headache days frequency compared to the baseline frequency. HIT-6 score reduction in each group after three months of treatment. The safety of treatment was evaluated by monitoring and documenting treatment-emergent adverse events (TEAE) in patients through regular follow-up procedures for three months. We will assess the phenotypic features of migraine.
  Interventions: Drug: Combined oral contraceptive
- the non-hormonal contraception group (Active Comparator): The arm will include 200 migraine patients diagnosed according to ICHD3-beta criteria. The patients are not receiving any hormonal contraception and will receive propranolol 80-160mg daily and ibuprofen 200-400 mg only in acute migraine attacks for 3 months. We will assess The change in migraine days per 28 days, the number of migraine days after three months of treatment, and the percentage of patients who achieved ≥ 50% reduction in the monthly headache days frequency compared to the baseline frequency. HIT-6 score reduction in each group after three months of treatment. The safety of treatment was evaluated by monitoring and documenting treatment-emergent adverse events (TEAE) in patients through regular follow-up procedures for three months. We will assess the phenotypic features of migraine.
  Interventions: Drug: Vaginal Ring

INTERVENTIONS:
Drug: Combined oral contraceptive — The arm will include 200 migraine patients diagnosed according to ICHD3-beta criteria. The patients are regular users of COCs and will receive propranolol 80-160mg daily and ibuprofen 200-400 mg only in acute migraine attacks for 3 months.
  Arms: the COCs group
Drug: Vaginal Ring — The arm will include 200 migraine patients diagnosed according to ICHD3-beta criteria. The patients are users of mechanical contraceptive methods and will receive propranolol 80-160mg daily and ibuprofen 200-400 mg only in acute migraine attacks for 3 months.
  Arms: the non-hormonal contraception group

SUMMARY:
The investigators will assess the effect of combined oral contraceptive pills (COCs) on migraine features and treatment response to allow better interpretation of the exact consequence of hormonal contraceptive use on migraineurs.

DETAILED DESCRIPTION:
The investigators will use a questionnaire to detect the migraineur demographic and clinical features (disease duration, attack frequency and duration, pain intensity assessed by visual analogic scale, HIT score in female patients on regular COCs

* Special emphasis was put on clinical phenotype (for example, the character of pain, location, associated symptoms, etc.); vascular risk factors (hypertension, diabetes, smoking); history of cerebrovascular events and other conditions (collagen disorders, hepatic disorders, blood diseases, heart, kidneys), and family history.
* All the patients will undergo clinical neurological and general physical examinations, and migraine history and associated phenotypic features will be established.

ELIGIBILITY:
Inclusion Criteria:

* female migraine patients on COCs or mechanical contraceptive methods, according to the International Classification of Headache Disorders 3rd edition, aged 18-55 years

Exclusion Criteria:

1. Patients with major neurological conditions such as (epilepsy, ischemic or hemorrhagic stroke, multiple sclerosis, mitochondrial diseases, and brain tumors).
2. pregnant, lactating, and menopausal patients.
3. Patients with any contraindications to ibuprofen or propranolol.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients who achieved ≥ 50% change in the monthly migraine days frequency compared to the baseline frequency | 90 days
  We will assess The percentage of patients who achieved ≥ 50% change in the monthly headache days frequency compared to the baseline frequency in each group

SECONDARY OUTCOMES:
The severity of migraine attack on VAS score after three months of treatment | 3 months
  After three months of treatment, the investigators will assess the severity of migraine attacks on VAS scores.
  VAS is a scale from one to ten where one is the least severe pain while ten is the most severest pain
HIT-6 score change in each group after three months of treatment | 3 months
  The investigators assessed the absolute change in HIT6 score, the Headache Impact Test-6 (HIT-6) assessed the burden of headache in each group; the HIT-6 consists of six items: pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress, the patient answers each of the six related questions using one of the following five responses: "never", "rarely", "sometimes", "very often," or "always." These responses are summed to produce a total HIT-6 score that ranges from 36 to 78, where a higher score indicates a greater impact of headache on the daily life of the respondent. It has four impact grades: little-to-no impact (HIT-6 score: 36-49), moderate impact (HIT-6 score: 50-55), substantial impact (HIT-6 score: 56-59), and severe impact (HIT-6 score: 60-78)
The monthly migraine days per month | 3 months
  The investigators will assess the change in migraine days per month in each group
The duration of migraine attack in hours after three months of treatment | 3 months
  After three months of treatment, the investigators will assess the duration of migraine attacks in hours in each group
percentage of phenotypic features after three months of treatment | 3 months
  After three months of treatment, the investigators will assess percentage of phenotypic features in each group.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafr Elsheikh University Hospital, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No
All the data supporting this research's findings may be available from Sherihan R.Ahmed, upon reasonable request

REFERENCES:
- [Result] Lipton RB, Scher AI, Kolodner K, Liberman J, Steiner TJ, Stewart WF. Migraine in the United States: epidemiology and patterns of health care use. Neurology. 2002 Mar 26;58(6):885-94. doi: 10.1212/wnl.58.6.885. PMID 11914403
- [Result] Lipton RB, Liberman JN, Kolodner KB, Bigal ME, Dowson A, Stewart WF. Migraine headache disability and health-related quality-of-life: a population-based case-control study from England. Cephalalgia. 2003 Jul;23(6):441-50. doi: 10.1046/j.1468-2982.2003.00546.x. PMID 12807523
- [Result] Mushet GR, Miller D, Clements B, Pait G, Gutterman DL. Impact of sumatriptan on workplace productivity, nonwork activities, and health-related quality of life among hospital employees with migraine. Headache. 1996 Mar;36(3):137-43. doi: 10.1046/j.1526-4610.1996.3603137.x. PMID 8984084